CLINICAL TRIAL: NCT00621569
Title: A Culturally Appropriate Intervention in Hypertensive African-Americans Based on the DASH Diet-The ADAPT Hypertension Study = Altering Diet for African American Populations to Treat Hypertension
Brief Title: ADAPT-Altering Diet for African American Populations to Treat Hypertension
Acronym: ADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jamy Ard, MD, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F0408110045; U01HL079171 (NIH)
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Hypertension
Keywords: Blood Pressure; Dash Diet
MeSH Terms: conditions — Hypertension | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Group intervention with no dietary focus
  Interventions: Behavioral: Intervention with no dietary component - information regarding useful life skills
- 2 (Experimental): DASH diet intervention
  Interventions: Behavioral: Dietary Approaches to Stop Hypertension-The DASH diet

INTERVENTIONS:
Behavioral: Dietary Approaches to Stop Hypertension-The DASH diet — The purpose of this study is to create a culturally appropriate diet to test the effectiveness of the intervention to lower blood pressure in a grou pof African American individuals at risk for developing hypertension (pre-hypertension) and those with mild hypertension (stage I).
  Arms: 2
Behavioral: Intervention with no dietary component - information regarding useful life skills — Participants receive information regarding useful life skills in a group setting
  Arms: 1

SUMMARY:
The purpose of the study is to develop a culturally appropriate DASH intervention and test the effectiveness of the intervention lower blood pressure in a group of African American participants at risk for developing hypertension (pre-hypertension) and those with mild hypertension (stage I).

DETAILED DESCRIPTION:
The effectiveness of the Dietary Approaches to Stop Hypertension (DASH) diet has shown to have limited impact on blood pressure control among African Americans, which might be explained by inappropriate adaptation to African American culture and tradition. Therefore, the adequate adaptation of the DASH diet would result in blood pressure control among African-Americans. Using the nominal group technique as a part of the formative assessment, this project proposes to identify key cultural variables that impact dietary patterns for African Americans. Based on those results, a modified behavioral intervention will be developed and tested in African Americans with pre-hypertension or stage I hypertension. Primary outcomes will include change in systolic and diastolic blood pressure at six months. It is expected that this project will contribute an additional tool for physicians, patients and health care systems to improve hypertension control amongst African Americans. The specific aims for this dietary intervention are: (1) to develop a modified DASH dietary pattern that is culturally appropriate for African-Americans by using principals of formative analysis and (2) to conduct a randomized, controlled trial to determine the effectiveness of the modified DASH dietary pattern in reducing blood pressure for a cohort of African-Americans with pre-hypertension or stage I hypertension to a usual care control group.

ELIGIBILITY:
Inclusion Criteria:

* Baseline SBP 120-159 mmHg and DBP 80-95 mmHg
* Age 25 or older as of the initial screening visit
* Willing and able to participate fully in all aspects of the intervention
* Not on rigid diet
* Provide informed consent
* BMI 18.5-45 kg/m2

Exclusion Criteria:

* Regular use of anti-hypertensive drugs or other drugs that raise or lower BP (any in previous three months)
* Current use of insulin or oral hypoglycemic agents
* Use of oral corticosteroids >5 days/month on average
* Current use of medications for treatment of psychosis or manic-depressive illness
* Use of oral breathing medications other than inhalers > 5 days/month on average
* Use of weight-loss medications in previous 3 months

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2005-01; Primary Completion 2008-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure with dietary intervention | 6 months

SECONDARY OUTCOMES:
Change in weight | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jamy D Ard, MD, Principal Investigator — University of Alabama at Birmingham; Catarina Kiefe, MD, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Department of Nutrition Sciences, Birmingham, Alabama, United States

REFERENCES:
- See also: Alabama Collaboration for Cardiovascular Equality (ACCE) is an initiative under the leadership of Drs. Catarina Kiefe and Sandral Hullett and is comprised of STORIES (NCT00101491), led by Dr. Thomas Houston, and ADAPT (NCT00621569), led by Dr. Jamy Ard — http://clinicaltrials.gov/show/NCT00101491